CLINICAL TRIAL: NCT04503291
Title: Comparison Between Transpapillary and Suprapapillary Metal Stent Placement With Endoscopic Sphincterotomy in Common Bile Duct Malignant Obstruction: Prospective Randomized Controlled Study
Brief Title: Comparison Between Transpapillary and Suprapapillary Metal Stent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bucheon St. Mary's Hospital (Other)
Collaborators: Seoul St. Mary's Hospital (Other); Incheon St.Mary's Hospital (Other); St Vincent's Hospital (Other)
Responsible Party: Principal Investigator, Jae Hyuck Chang, Professor, Bucheon St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BucheonStMarys
Record Dates: First submitted 2020-07-30; First posted 2020-08-07 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Common Bile Duct Stricture
Keywords: metal stent; common bile duct obstruction; endoscopic retrograde cholangiopancreatography

STUDY DESIGN:
Intervention Model Description: 1. supra-papillary metal stent group
  2. trans-papillary metal stent group
Who Masked: Participant, Outcomes Assessor
Masking Description: Assigned groups are secreted to the participant and outcome assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supra-papillary metal stent group (Experimental): The distal ends of metal stents are located above the major papilla in the common bile duct.
  Interventions: Procedure: Metal stent placement
- trans-papillary metal stent group (Active Comparator): The distal ends of metal stents are located below the major papilla in the duodenum.
  Interventions: Procedure: Metal stent placement

INTERVENTIONS:
Procedure: Metal stent placement — Non-covered biliary metal stents are placed by endoscopy. The distal ends of metal stents are located above the major ampulla in the common bile duct or below the major ampulla in the duodenum.

SUMMARY:
If surgical treatment is not possible in patients with malignant obstruction in the common bile duct, placing metal stents using endoscopy is a standardized treatment to resolve biliary obstruction. The metal stent is located in the bile duct to cover the stenotic portion by malignant tumors.

The lower end of the metal stent can be located inside the common bile duct above the major ampulla or in the duodenum through the major ampulla. These two procedures with supra- or trans-papillary stents are currently being performed in general clinical practices, depending on the preference of the endoscopists. Until now, the comparison of the clinical results of the two procedures has been scarcely studied, and there is no prospective study yet. Therefore, researchers aim to compare the clinical results of two stent procedures through prospective randomized controlled studies.

DETAILED DESCRIPTION:
If surgical treatment is not possible in patients with malignant obstruction in the common bile duct, endoscopic metal stent placement to resolve biliary obstruction is a standard treatment that is commonly performed. The metal stents relieve the bile duct stenosis by malignant tumors, helping to drain the bile and improving jaundice. There is no doubt that the center of the metal stent is located in the central part of the biliary stricture, but the location of the lower end of the metal stent is not fixed. The lower end of the metal stent can be located in two main locations, either in the common bile duct above the major ampulla or in the duodenum through the major ampulla. These procedures with supra- or trans-papillary stents are performed in common and are determined by the operator's preference.

According to several retrospective studies so far, trans-papillary metal stents were effective in improving the initial biliary obstruction, but there was no difference in their long-term effects. Mao et al. showed that trans-papillary metal stents increase jaundice-free survival, and Shin et al. revealed the advantages of trans-papillary metal stents because they had a high success rate of secondary endoscopic procedures. On the contrary, Okamoto et al. showed that acute cholangitis more developed after trans-papillary metal stents placement, while Joe et al. revealed the advantages of supra-papillary metal stents because they reduce acute pancreatitis after the procedures. It has not yet been determined which method is effective. So far studies are all retrospective, and some of them placed the metal stents in a percutaneous way rather than endoscopy without sphincterotomy. Besides, some studies included intra-hepatic or hilar bile duct strictures, making it difficult to interpret the results.

Therefore, through a prospective randomized controlled study, the researchers want to compare the clinical results of supra- and trans-papillary metal stents placed by endoscopes in malignant common bile duct obstruction.

ELIGIBILITY:
Inclusion Criteria:

* patients with common bile duct obstruction due to malignancy

Exclusion Criteria:

* intrahepatic or perihilar bile duct obstruction (except Klatskin type I)
* patients who have operability or want surgery
* strictures located within 2 cm from the end of distal common bile duct
* patients who are not able to undergo endoscopy due to cardiovascular or pulmonary diseases
* patients whose informed consents are not received
* patients in whom an endoscope can not access to the ampulla due to anatomical deformity by previous surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-12 (Estimated)

PRIMARY OUTCOMES:
Stent function maintenance duration | through study completion, an average of 1 year
  jaundice free survival

SECONDARY OUTCOMES:
stone or sludge occurrence | through study completion, an average of 1 year
  in-stent or above stent bile duct stone formation
in-stent stenosis or tumor overgrowth | through study completion, an average of 1 year
  stenosis due to tumor growth: in-stent or over the stent
acute cholangitis occurrence | through study completion, an average of 1 year
  after procedure acute cholangitis occurrence rate
stent migration rate | through study completion, an average of 1 year
  spontaneous migration rate
overall survival | From date of randomization until the date of date of death from any cause, assessed up to 36 months
  duration between stent placement and death

CONTACTS AND LOCATIONS:
Locations (1):
- Jae Hyuck Chang, Bucheon-si, Kyunggi, South Korea

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date
Access Criteria: * Investigators whose proposed use of the data has been approved by an independent review committee
  * To achieve aims in the approved proposal
  * Proposals may be submitted up to 36 months following article publication.